CLINICAL TRIAL: NCT03454971
Title: Multidisciplinary Consultation at the GHM Hospital of Grenoble (France) for the Establishment of an Oral Anti-cancer Drug Therapy : Feasibility, Security, and Evaluation of Patients' and City Health Professionals' Satisfaction.
Brief Title: Health Course of Patients Undergoing Per os Anti-cancer Therapy.
Acronym: MinOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018/01-CGT-GHMG
Record Dates: First submitted 2018-02-05; First posted 2018-03-06 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MinOS arm (Experimental): Patients are followed according to MinOS protocol:
  Interventions: Other: MinOS protocol

INTERVENTIONS:
Other: MinOS protocol — At Day 1, Cycle 1 and 2 of the patient's oral therapy :
  * Consultation with a hospital pharmacist
  * Consultation with a nurse care coordinator
  * Consultation with the patient's oncologist/hematologist
  During this multidisciplinary consultation, will be reviewed :
  * potential medical interactions,
  * possible adverse effects of therapy,
  * information on the prescribed drug,
  * informations on the patient's lifestyle, ...
  At day 8 and 15, cycle 1 and 2 :
  Phone call from the nurse care coordinator during which will be reported the adverse effects and adherence issues. If needed, the nurse care coordinator can provide complementary information about the treatment.
  The MINOS protocol follow up will end with a consultation with the patient's oncologist/hematologist, at day 1 cycle 3.

SUMMARY:
During the last few years, the medical care of oncohematologic cancers diagnosed patients was shaken by the arrival of new therapies : targeted therapies. Very efficient, these therapies use the oral pathway in most cases, and are taken at home. These treatments show plenty of drug interactions and side effects aren't rare and require, in their own, a rigorous follow up in order to reduce their occurrence, intensity and their impact on patients' quality of life. A bad management of the treatment could lead to an inacceptable toxicity, or to its premature interruption.

With all the new administration and follow up strains in mind, we want to elaborate the medical pathway structure for these patients by reinforcing the nurse coordination and by integrating another healthcare professional : the hospital pharmacist, which is a professional especially implicated in the drug delivery, the control of drug interactions and medical advices relative to the given drug.

Private healthcare professionals (referring physicians, pharmacists, private nurses), unsufficiently trained and informed about these new treatments and their side effects, are asking for further information concerning the drugs prescribed to their patients, and are willing to keep open a communication line for the home follow up.

These patients, who are autonomously taking their medication, are in need to be informed and supported to insure the good management of the drug, while taking in account their environment, their knowledge of their cancer and treatment and also of all the issues that could occur during their therapy, in order to resolve them.

We propose a multidisciplinary medical care taking place at the very beginning of an oral therapy treatment, in order to ensure the security of the drug administration. Patients and healthcare professionals will be closely followed during the first two treatment cycles. After this, side-effects incidence are less frequent and the usual oncohematologic follow up is sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Patient who treated at the Groupe Hospitalier Mutualiste for an oncohematological pathology, and for which targeted oral therapy is indicated (Tarceva, Afinitor, Sutent, Ibrance, Revlimid, Zydelig, Imbruvica)
* Patient who has given its written consent
* Patient affiliated or beneficiary of social security system

Exclusion Criteria:

* ECOG performance score < 2
* Patient already included in an interventional clinical research protocol
* Patients protected by French law from clinical research inclusion (pregnant, in labour, breastfeeding, legally protected, under judiciary or administrative liberty deprivation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Number of patients that followed the entirety of MinOS follow-up. | At the eighth follow-up, which is 8 weeks from baseline, except for Sutent treatment (12 weeks from baseline)
  - 91% of included patients must have followed the entirety of MinOS follow up. A patient has followed the entirety of MinOS follow up only if he has attended to each and every one of their 8 scheduled follow up (4 phone calls + 4 consultations)

SECONDARY OUTCOMES:
Toxicity evaluation of targeted oral therapies | Day 8 and 15 of 1st treatment cycle ; Day 1, 8 and 15 of 2nd treatment cycle ; Day 1 of 3rd treatment cycle. One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
  - toxicity nature and grade according to CTCAE classification.
Evaluation of observance | End of the 1st and 2nd treatment cycle. One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
  - Observance score of Morisky
Number of unscheduled phone calls | At the end of the 2nd cycle. One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
Number of unscheduled hospitalizations | At the end of the 2nd cycle. One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
Number of private healthcare professionals visit | At the end of the 2nd cycle. One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
Number of private healthcare professionals' phone call to the hospital | At the end of the 2nd cycle. One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
Description of the exchange of information between the hospital and independent health professionals | Day 1 of the 1st and 2nd treatment cycles. One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
  - Evaluation of the utilization of "patients-files": Patients will be asked whether they make use of their "patient-files" and whether they share them with their healthcare professionals, if needed. (YES/NO)
Description of the patient's independence in regard of his treatment and pathology | At the end of the 2nd cycle. One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
  - Number of patient's phone call to the hospital
Evaluation of patient's satisfaction in regard of MinOS protocol | At the end of the patient's therapy within MinOS framework (end of cycle 2). One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
  - Satisfaction survey answered by patients
Evaluation of private healthcare professionals' satisfaction in regard of MinOS protocol | At the end of the patient's therapy within MinOS framework (end of cycle 2). One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
  - Satisfaction survey answered by private healthcare professionals
Evaluation of the quality of life for patients recruited in MinOS protocol | Day 1 of 1st, 2nd and 3rd cycle of treatment. One treatment cycle = 4 weeks, except for Sutent treatment: 1 cycle = 6 weeks
  - Score of QLQ-C30 questionnaire
Number of concomitant drug prescription modification by the hospital pharmacist due to drug interactions with the cancer treatment | At the end of the 2nd cycle. One treatment cycle = 4 weeks, except for Sutent treatment : 1 cycle = 6 weeks
  - A high number of prescription modification will mean an important part played by the hospital pharmacist, whereas a low number of modification will mean that adding a hospital pharmacist consultation to the standard care isn't relevant.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Mutualiste de Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu G, Franssen E, Fitch MI, Warner E. Patient preferences for oral versus intravenous palliative chemotherapy. J Clin Oncol. 1997 Jan;15(1):110-5. doi: 10.1200/JCO.1997.15.1.110. PMID 8996131
- [Background] Noens L, van Lierde MA, De Bock R, Verhoef G, Zachee P, Berneman Z, Martiat P, Mineur P, Van Eygen K, MacDonald K, De Geest S, Albrecht T, Abraham I. Prevalence, determinants, and outcomes of nonadherence to imatinib therapy in patients with chronic myeloid leukemia: the ADAGIO study. Blood. 2009 May 28;113(22):5401-11. doi: 10.1182/blood-2008-12-196543. Epub 2009 Apr 6. PMID 19349618
- [Background] Eliasson L, Clifford S, Barber N, Marin D. Exploring chronic myeloid leukemia patients' reasons for not adhering to the oral anticancer drug imatinib as prescribed. Leuk Res. 2011 May;35(5):626-30. doi: 10.1016/j.leukres.2010.10.017. Epub 2010 Nov 20. PMID 21095002
- [Background] Compaci G, Ysebaert L, Oberic L, Derumeaux H, Laurent G. Effectiveness of telephone support during chemotherapy in patients with diffuse large B cell lymphoma: the Ambulatory Medical Assistance (AMA) experience. Int J Nurs Stud. 2011 Aug;48(8):926-32. doi: 10.1016/j.ijnurstu.2011.01.008. Epub 2011 Feb 23. PMID 21349519
- [Background] Compaci G, Rueter M, Lamy S, Oberic L, Recher C, Lapeyre-Mestre M, Laurent G, Despas F. Ambulatory Medical Assistance--After Cancer (AMA-AC): A model for an early trajectory survivorship survey of lymphoma patients treated with anthracycline-based chemotherapy. BMC Cancer. 2015 Oct 24;15:781. doi: 10.1186/s12885-015-1815-7. PMID 26498342
- See also: [Cancer National Institut. Plan Cancer 2014-2019] (French). Febr 2015. — http://www.e-cancer.fr/Expertises-et-publications/Catalogue-des-publications/Plan-Cancer-2014-2019
- See also: [Oncorif. White book : Organisation and care of patient undergoing oral targeted therapy in hematology] (french). Nov 2016. — http://www.oncorif.fr/wp-content/uploads/2017/06/Livre_Blanc_Hemopathies_malignes-_Version_Numerique_Nov_16.pdf
- See also: [Cancer National Institut. Hematology : adverse effects of anti-cancer oral therapies] (french). Sept 2014. — https://www.af3m.org/uploads/PDF/Actualites/anticancereux_oraux_-_effets_indesirables_-_enquete_patients_-_ete_2014.pdf
- See also: [APM. Oral chemotherapies : nurses' part and role] (french). July 2014. — http://www.infirmiers.com/profession-infirmiere/cooperations-interprofessionnelles/chimiotherapies-orales-place-des-infirmieres.html
- See also: ATHOS team (french) — http://hopitaux-paris-centre.aphp.fr/cancerologie/
- See also: [Cancer National Institut. oral anti-cancer therapy patients medical course : referral] (french). Nov 2016. — http://www.e-cancer.fr/Expertises-et-publications/Catalogue-des-publications/Parcours-de-soins-d-un-patient-traite-par-anticancereux-oraux-Reponse-saisine
- See also: [Cancer National Institut. Cancer Plan from 2003 to 2007] (french) — http://www.e-cancer.fr/Plan-cancer/Les-Plans-cancer-de-2003-a-2013/Le-Plan-cancer-2003-2007
- See also: [Cancer National Institut. Cancer Plan from 2009 to 2013] (french) — http://www.e-cancer.fr/Plan-cancer/Les-Plans-cancer-de-2003-a-2013/Le-Plan-cancer-2009-2013
- See also: [Cancer National Institut. Cancer Plan from 2014 to 2019] (french) — http://www.e-cancer.fr/Plan-cancer/Plan-cancer-2014-2019-priorites-et-objectifs